CLINICAL TRIAL: NCT01920425
Title: Kinesia HomeView - Home Diary Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1311DH; 1311DH (Other: Great Lakes NeuroTechnologies)
Record Dates: First submitted 2013-08-07; First posted 2013-08-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; dyskinesia; fluctuations; tremor; bradykinesia; levodopa
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Tremor; Hypokinesia

ARMS (2):
- Hand-written diary first (Other): Participants in this group will use the hand-written diary for the first two week and switch to Kinesia HomeView and the electronic diary for the second two weeks.
  Interventions: Device: Kinesia HomeView; Other: Hand-written diary
- Kinesia HomeView first (Other): Participants in this group will use Kinesia HomeView and the electronic diary for the first two week and switch to the hand-written diary for the second two weeks.
  Interventions: Device: Kinesia HomeView; Other: Hand-written diary

INTERVENTIONS:
Device: Kinesia HomeView — Motion sensor based telemedicine system for assessment of movement disorder motor symptoms in the home. Includes automated motor assessment using motion sensor and electronic dyskinesia diary.
Other: Hand-written diary — Hand-written paper diary indicating state (Off, On without dyskinesias, on with non-troublesome dyskinesias, on with troublesome dyskinesias) at 30 minute intervals.

SUMMARY:
The objective is to compare the sensitivity and test-retest reliability of Kinesia HomeView to electronic and hand-written diaries for tracking medication state in the home. Demonstrating comparable or superior results will further support use of the Kinesia HomeView system as an outcome measure in clinical drug trials.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* On a stable antiparkinsonian medication regimen that includes levodopa for at least 4 weeks
* Experiencing dyskinesia more than 25% of the waking day (score ≥ 2 on Unified Parkinson's Disease Rating Scale item 32)
* With dyskinesias at least moderately disabling (score ≥ 2 on Unified Parkinson's Disease Rating Scale item 33)
* Capable of accurately completing diaries
* Capable of accurately using Kinesia HomeView

Exclusion Criteria:

* Significant medical or psychiatric illness
* Subjects not capable of following the required clinical instructions
* Serious medical conditions that would compromise safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Test-retest reliability | 4 weeks
  Test-retest reliability will be compared between Kinesia HomeView measures, hand-written diary entries, and electronic diary entries.

SECONDARY OUTCOMES:
Kinesia HomeView usability questionnaire | After 4 weeks
  Questionnaires on the usability of Kinesia HomeView will be completed following the 4-week data collection period.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies Inc.
Locations (1):
- Great Lakes NeuroTechnologies Inc, Valley View, Ohio, United States